CLINICAL TRIAL: NCT06179706
Title: 11C-choline PET/CT Based Helical Tomotherapy as Innovative Treratment Approach for Bone Metastases in Prostate Cancer Patients.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: Colina-osso
Record Dates: First submitted 2023-11-30; First posted 2023-12-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 11C-choline PET/CT — In our study we evaluated the efficacy of high-dose RT guided by 11C-Choline PET/CT on bone metastases in prostate cancer patients with a limited number of metastases.

SUMMARY:
The number of metastases may reflect the biological aggressiveness of the tumor and may determine the possibility of performing potential curative interventions such as surgery or high-dose targeted radiotherapy (RT). Until a few years ago, the treatment of choice for metastatic prostate cancer was androgen deprivation (TDA). This treatment was carried out as palliative care in order to postpone the progression of the disease or reduce symptoms. Patients with prostate cancer with a limited number of metastases, similarly to patients suffering from other solid tumors, can be considered as patients with disease that has limited capacity to cause further secondary effects. In this scenario, the primary treatment in patients with carcinoma localized prostate, is characterized by radical prostatectomy, followed by measurement of prostate specific antigen (PSA) during follow-up. After primary prostatectomy, PSA values > 0.2 ng/mL are indicative of disease recurrence, but it is not possible to determine whether the recurrence is local or distant. Furthermore, imaging modalities, such as bone scanning and computed tomography (CT), do not have sufficient sensitivity to detect the presence of metastatic disease in patients with low PSA levels. Positron emission tomography/CT with 11C-choline is able to detect local or distant metastases with a sensitivity and specificity greater than 85% in patients with biochemical disease recurrence. 11C-Choline PET/CT can be a valid tool both for diagnosis and for guiding radiotherapy treatments in these patients for whom it is not possible to obtain a definitive diagnosis with conventional diagnostic procedures. There are currently few studies that have described the use of 11C-choline PET/CT to guide treatment for bone metastases; the limitations of these studies concern the small number of patients and the short follow-up. The aim of this retrospective observational study was to evaluate the efficacy of 11C-choline PET/CT as a guide to the treatment of helical tomotherapy for an innovative therapeutic approach in bone metastases in a population of patients affected by prostate cancer with a limited number of metastasis.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with less than 3 bone lesions found on C11-Choline PET/CT
* availability of clinical follow-up using serial PSA assays.

Exclusion Criteria:

<18 years patients

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: patients suffering from prostate cancer who have undergone primary curative treatment and who have presented biochemical recurrence of the disease.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
11C-choline PET/CT to the treatment of patients with prostate cancer with a limited number of metastasis. | 1 year
  Retrospective observational study with 11C-choline PET/CT for the treatment of helical tomotherapy for an innovative therapeutic approach in bone metastases in a population of patients affected by prostate cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No